CLINICAL TRIAL: NCT03890835
Title: Comparative Evaluation of Postoperative Pain and Success Rate After Pulpotomy in Mature Permanent Molars Using Biodentine Versus Mineral Trioxide Aggregate (MTA) as Capping Materials: A Randomized Clinical Trial
Brief Title: Pulpotomy in Mature Permanent Molars Using Biodentine Versus MTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youssef Andraws, Postgraduate Student, Department of Endodontics, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-03-10
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Pulpotomy; Mineral Trioxide Aggregate (MTA); Biodentine; Vital pulp therapy; Postoperative pain; Overall success
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Type: Two arm, parallel, randomized clinical trial. Allocation ratio: 1:1 Framework: Superiority.
Who Masked: Participant
Masking Description: The study will be participant-blind where the participant will not know the intervention done.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral Trioxide Aggregate (MTA) (Active Comparator)
  Interventions: Procedure: MTA Pulpotomy.
- Biodentine (Experimental)
  Interventions: Procedure: Biodentine Pulpotomy

INTERVENTIONS:
Procedure: MTA Pulpotomy. — Pulpotomy using MTA.
  Arms: Mineral Trioxide Aggregate (MTA)
Procedure: Biodentine Pulpotomy — Pulpotomy using Biodentine
  Arms: Biodentine

SUMMARY:
The aim of this study is to compare treatment outcomes of pulpotomy in mature permanent teeth using Biodentine versus MTA regarding postoperative pain and success rate.

DETAILED DESCRIPTION:
* Patients will be clinically and radiographically examined and their eligibility will be assessed.
* Eligible patients will be randomly assigned to one of 2 groups: experimental group (pulpotomy using Biodentine) and the control group (pulpotomy using MTA).
* After adminsrtation of local anesthesia, pulpotomy will be done under rubber dam isolation. The pulp tissue will be removed until the level of the orifices of the canals. After hemostasis is achieved, the capping material will be placed. In the experimental group, the capping material is Biodentine while in the control group, the capping material is MTA
* The cavities will be sealed with resin-modified glass ionomer. Then the teeth will be permanently restored with composite . A post-operative radiograph will be taken.
* The patients will be given a pain diary based on Numerical Rating Scale (NRS) and asked to rate their pain level at the specified times.
* The patients will be recalled after 6 and 12 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging between 18-40 years old
* Patients with symptomatic irreversible pulpitis.
* Radiographically: Absence or slight widening in periodontal ligament space.
* Systemically- healthy patients (ASA I or II).
* Patients who agree to attend for recall appointments and provide written consent.

Exclusion Criteria:

* Severe marginal periodontitis.
* Necrotic pulp, pulp polyp, tooth tender to percussion, clinical progression into periapical abscess, fistula.
* Non-restorable teeth, teeth with internal/external root resorption or root canal calcification.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain after 6 hours postoperatively | 6 hours postoperatively
  Each patient will be given a pain diary based on Numerical Rating Scale(NRS). NRS is an 11-point scale consisting of numbers from 0 through 10.
  0 reading represents "no pain"
  1- 3 readings represent "mild pain"
  4- 6 readings represent "moderate pain"
  7- 10 readings represent "severe pain"
Postoperative pain after 12 hours postoperatively | 12 hours postoperatively
  Each patient will be given a pain diary based on Numerical Rating Scale(NRS). NRS is an 11-point scale consisting of numbers from 0 through 10.
  0 reading represents "no pain"
  1- 3 readings represent "mild pain"
  4- 6 readings represent "moderate pain"
  7- 10 readings represent "severe pain"
Postoperative pain after 24 hours postoperatively | 24 hours postoperatively
  Each patient will be given a pain diary based on Numerical Rating Scale(NRS). NRS is an 11-point scale consisting of numbers from 0 through 10.
  0 reading represents "no pain"
  1- 3 readings represent "mild pain"
  4- 6 readings represent "moderate pain"
  7- 10 readings represent "severe pain"

SECONDARY OUTCOMES:
Overall (clinical and radiographic) success after 6 months postoperatively. | 6 months postoperatively
  Outcome of overall success will be determined based on clinical and radiographic examination. If there is either clinical or radiographic failure , then the case will be considered as an overall failure.
Overall (clinical and radiographic) success after 12 months postoperatively. | 12 months postoperatively
  Outcome of overall success will be determined based on clinical and radiographic examination. If there is either clinical or radiographic failure , then the case will be considered as an overall failure.

CONTACTS AND LOCATIONS:
Overall Officials: Youssef A. Kamal Elalfy, B.D.S., Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asgary S, Eghbal MJ, Fazlyab M, Baghban AA, Ghoddusi J. Five-year results of vital pulp therapy in permanent molars with irreversible pulpitis: a non-inferiority multicenter randomized clinical trial. Clin Oral Investig. 2015 Mar;19(2):335-41. doi: 10.1007/s00784-014-1244-z. Epub 2014 Apr 27. PMID 24771228
- [Background] Galani M, Tewari S, Sangwan P, Mittal S, Kumar V, Duhan J. Comparative Evaluation of Postoperative Pain and Success Rate after Pulpotomy and Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial. J Endod. 2017 Dec;43(12):1953-1962. doi: 10.1016/j.joen.2017.08.007. Epub 2017 Oct 20. PMID 29061359
- [Background] Bakhtiar H, Nekoofar MH, Aminishakib P, Abedi F, Naghi Moosavi F, Esnaashari E, Azizi A, Esmailian S, Ellini MR, Mesgarzadeh V, Sezavar M, About I. Human Pulp Responses to Partial Pulpotomy Treatment with TheraCal as Compared with Biodentine and ProRoot MTA: A Clinical Trial. J Endod. 2017 Nov;43(11):1786-1791. doi: 10.1016/j.joen.2017.06.025. Epub 2017 Aug 16. PMID 28822566